CLINICAL TRIAL: NCT03000881
Title: Evaluation of the Influence of Output on Skin Covered by Adhesives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP265_06
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohort 6 (Experimental): This is a sub-study testing the effect of real output applied under two adhesive strips after 8 hours.
  Interventions: Other: standard adhesive; Other: New adhesive strip

INTERVENTIONS:
Other: standard adhesive — This is a standard adhesive (hydrocolloid)
Other: New adhesive strip — This is a newly developed adhesive strip

SUMMARY:
The study investigates the impact real output has on peristomal skin covered by two different adhesives

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent
* Be at least 18 years of age and have full legal capacity
* Have had an ileostomy for more than one year
* Have intact skin on the area used in the evaluation
* Has an ileostomy with a diameter up to 35 mm
* Have a peristomal area accessible for application of adhesive strips

Exclusion Criteria:

* Currently receiving or have within the past 2 month received radio- and/or chemotherapy
* Currently receiving or have within the past month received topical steroid treatment in the peristomal skin area or systemic steroid (tablet/injection) treatment.
* Are pregnant or breastfeeding
* Having dermatological problems in the peristomal- or abdominal area (assessed by investigating scientist)
* Participating in other interventional clinical investigations or have previously participated in this evaluation -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Trans Epidermal Water Loss | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lene F Nielsen, M. Sc, Principal Investigator — Head of preclinical department
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No